CLINICAL TRIAL: NCT04628468
Title: Patient Reported Outcome of Rehabilitation and Quality of Life in Computer Literate Patients Undergoing Primary Knee or Hip Arthroplasty and Randomized to Rehabilitation With or Without the Possible Use of a Mobile Application.
Brief Title: Patient Reported Outcome Measures (PROMs) in Rehabilitation With or Without the Possible Use of a Mobile Application After Primary Knee or Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: National Institute for Health and Disability Insurance (NIHDI), Belgium (Unknown); Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCE HTA C2020-1
Record Dates: First submitted 2020-10-27; First posted 2020-11-13 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Arthroplasty, Replacement, Knee; Rehabilitation; Hip Arthrosis
Keywords: mobile application; patient reported outcomes, PROMs; physiotherapy; telerehabilitation
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Possibility to use the mobile application without a predefined number of physiotherapy sessions (Experimental): Rehabilitation after hip or knee arthroplasty with the option to use a mobile application and no predefined traditional physiotherapy.
  Interventions: Device: moveUp
- Possibility to use the mobile application with a predefined number of physiotherapy sessions (Experimental): Rehabilitation after hip or knee arthroplasty with the option to use a mobile application and a predefined number of traditional physiotherapy sessions
  Interventions: Device: moveUp; Other: Predefined number of traditional physiotherapy sessions
- Usual care (No Intervention): Rehabilitation after hip or knee arthroplasty without the use of a mobile application.

INTERVENTIONS:
Device: moveUp — Mobile application for use in the rehabilitation of primary knee and hip arthroplasty
  Arms: Possibility to use the mobile application with a predefined number of physiotherapy sessions; Possibility to use the mobile application without a predefined number of physiotherapy sessions
Other: Predefined number of traditional physiotherapy sessions — exercises with a physiotherapist being physically present
  Arms: Possibility to use the mobile application with a predefined number of physiotherapy sessions

SUMMARY:
Rehabilitation after primary knee or hip arthroplasty may include performing exercises with a physiotherapist. For patients who can work well with a computer, tablet or smartphone, it is now possible to use a mobile application (e.g. moveUp) to carry out a large part of the exercises more independently. This is done with online guidance by a physiotherapist via a mobile application that is CE marked in Europe.

This study will investigate whether the effect of the mobile application on knee or hip rehabilitation and quality of life is equal to that of standard care (i.e. without the use of a mobile application).

DETAILED DESCRIPTION:
Via the moveUP Coach App, patients receive personalized rehabilitation for knee or hip replacement, both before and after surgery. This mobile application is on the market, meets the legal requirements in Europe and has been provisionally remunerated under an agreement (convention) between the mandatory health insurance (NIHDI) and the hospital that participate in this study.

Eligible patients will be randomized to one of the three treatment options of the study:

1. The "usual care group" will not be informed in detail about the mobile application and will receive usual rehabilitation care for knee- or hip replacement.
2. The group "possibility to use the mobile application with a predefined number of physiotherapy sessions" will receive all necessary information on the mobile application and can still decide whether or not to receive rehabilitation with online guidance by a physiotherapist via the mobile application. A predefined number of traditional physiotherapy sessions is combined with the use of the mobile app in this group.
3. The group "possibility to use the mobile application without a predetermined number of physiotherapy sessions" will receive all necessary information on the mobile application and can still decide whether or not to receive rehabilitation with online guidance by a physiotherapist via the mobile application. No predefined number of traditional physiotherapy sessions are required.

The patient will be asked to complete 2 questionnaires (KOOS-JR/HOOS-JR and EQ5D-5L) at baseline, 6 weeks and 6 months after arthroplasty. These patient reported outcomes will give an indication on the rehabilitation outcome and quality of life compared in the 3 groups.

At the end of the study, a health economic evaluation is foreseen by the Federal Knowledge Center for Healthcare (KCE). In this way the results can be helpful in getting a more definitive refund for the mobile application in Belgium.

ELIGIBILITY:
Eligibility criteria:

1. The patient is aged 18 years or older, has a Belgian National Number, is insured by a Belgian sickness fund, and is not staying in a nursing home or long term rehabilitation centre.
2. The patient has sufficient knowledge of Dutch, French, German or English.
3. The patient has a planned date between the next 1 to 8 weeks for a primary unilateral unicompartmental knee arthroplasty (UKA); a bicompartmental knee arthroplasty, (BKA), consisting of either two UKA or a UKA and a patellar replacement; or a total knee arthroplasty (TKA) or a total hip arthroplasty (THA).
4. The patient is not planned to have a peri-operative procedure (e.g. intra-articular catheter) or postoperative procedure that is expected to significantly impact the rehabilitation in and out of hospital.
5. In the 6 months after arthroplasty the patient is not planned to have surgery that may impact the arthroplasty rehabilitation.
6. The patient is not suffering from a medical condition (e.g. Parkinson, multiple sclerosis, cerebrovascular accident) that is expected to significantly impact the rehabilitation or that constitutes a contra-indication for the use of the mobile application.
7. The patient confirms to have easy and daily access to the internet, a mobile phone, a personal email address and a computer, tablet or smartphone, until 8 months after randomization.
8. The patient does not upfront exclude the possibility whereby part of the rehabilitation is performed without a physical therapist physically being present.
9. The patient is willing to complete online the patient reported outcomes and is aware that if he/she fails in this computer literacy test (performed before randomization) he/she will not be randomized and hence not included in the study. He/she will receive usual rehabilitation care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Rehabilitation result 6 months after knee arthroplasty | 6 months after arthroplasty
  Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS-JR score). KOOS-JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Rehabilitation result 6 months after hip arthroplasty | 6 months after arthroplasty
  Hip dysfunction and Osteoarthritis Outcome score for Joint Replacement (HOOS-JR score). HOOS-JR is scored by summing the raw response (range 0-24) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.

SECONDARY OUTCOMES:
Rehabilitation result 6 weeks after knee arthroplasty | 6 weeks after arthroplasty
  Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS-JR score). KOOS-JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Rehabilitation result 6 weeks after hip arthroplasty | 6 weeks after arthroplasty
  Hip dysfunction and Osteoarthritis Outcome score for Joint Replacement (HOOS-JR score). HOOS-JR is scored by summing the raw response (range 0-24) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.
Quality of life assessment 6 weeks after arthroplasty | 6 weeks after arthroplasty
  EQ5D-5L score. This score describes and values health-related quality of life and consist (1) the EQ-5D descriptive system with 5 dimensions each having 5 response levels from 1 indicating no problems to 5 indicating extreme problems, and (2) the EQ visual analogue scale (EQ VAS), a 0-100 scale with 0 score the worst health the patient can imagine and 100 the best health the patient can imagine.
Quality of life assessment 6 months after arthroplasty | 6 months after arthroplasty
  EQ5D-5L score. This score describes and values health-related quality of life and consist (1) the EQ-5D descriptive system with 5 dimensions each having 5 response levels from 1 indicating no problems to 5 indicating extreme problems, and (2) the EQ visual analogue scale (EQ VAS), a 0-100 scale with 0 score the worst health the patient can imagine and 100 the best health the patient can imagine.

OTHER OUTCOMES:
Incidents | baseline until 6 months after arthroplasty
  Any malfunction or deterioration in the characteristics and/or performance of the medical device app, as well as any inadequacy in the labeling or the instructions for use which, directly or indirectly, might lead to or might have led to the death of a patient, or user or of other persons or to a serious deterioration in their state of health.
Sensitivity endpoint KOOS-JR at 6 weeks | baseline until 6 weeks after arthroplasty
  Change in KOOS-JR score from baseline at 6 weeks after arthroplasty. KOOS-JR is a Knee injury and Osteoarthritis Outcome Score for Joint Replacement. KOOS-JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Sensitivity endpoint HOOS-JR at 6 weeks | baseline until 6 weeks after arthroplasty
  change in HOOS-JR score from baseline at 6 weeks after arthroplasty. HOOS-JR is a Hip dysfunction and Osteoarthritis Outcome score for Joint Replacement. HOOS-JR is scored by summing the raw response (range 0-24) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.
Sensitivity endpoint EQ5D-5L at 6 weeks | baseline until 6 weeks after arthroplasty
  change in EQ5D-5L score from baseline at 6 weeks after arthroplasty. This score describes and values health-related quality of life and consist (1) the EQ-5D descriptive system with 5 dimensions each having 5 response levels from 1 indicating no problems to 5 indicating extreme problems, and (2) the EQ visual analogue scale (EQ VAS), a 0-100 scale with 0 score the worst health the patient can imagine and 100 the best health the patient can imagine.
Sensitivity endpoint KOOS-JR at 6 months | baseline until 6 months after arthroplasty
  Change in KOOS-JR score from baseline at 6 months after arthroplasty. KOOS-JR is aKnee injury and Osteoarthritis Outcome Score for Joint Replacement. KOOS-JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Sensitivity endpoint HOOS-JR at 6 months | baseline until 6 months after arthroplasty
  Change in HOOS-JR score from baseline at 6 months after arthroplasty. HOOS-JR is a Hip dysfunction and Osteoarthritis Outcome score for Joint Replacement. HOOS-JR is scored by summing the raw response (range 0-24) and then converting it to an interval score using a table provided. The interval score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.
Sensitivity endpoint EQ5D-5L at 6 months | baseline until 6 months after arthroplasty
  change in EQ5D-5L score from baseline at 6 months after arthroplasty. This score describes and values health-related quality of life and consist (1) the EQ-5D descriptive system with 5 dimensions each having 5 response levels from 1 indicating no problems to 5 indicating extreme problems, and (2) the EQ visual analogue scale (EQ VAS), a 0-100 scale with 0 score the worst health the patient can imagine and 100 the best health the patient can imagine.
Deaths | baseline until 6 months after arthroplasty
  anticipated and unanticipated deaths

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Van Der Straeten, Professor, Study Director — Health, Innovation and Research Institute UZ Ghent
Locations (11):
- Belgium (11):
  - Antwerp University Hospital, Antwerp
  - Centre Hospitalier Interrégional Edith Cavell (CHIREC), site Delta, Auderghem
  - Centre Hospitalier Interrégional Edith Cavell (CHIREC), Hôpital de Braine L'Alleud-Waterloo, Braine-l'Alleud
  - AZ Sint-Jan Brugge, Bruges
  - AZ Monica Deurne, Deurne
  - AZ Alma Eeklo, Eeklo
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Jan Yperman Ziekenhuis, Ieper
  - CHU de Liège, site du Sart Tilman, Liège
  - AZ Damiaan, Ostend

IPD SHARING:
Plan to Share IPD: No